CLINICAL TRIAL: NCT02339545
Title: Coronary Flow Reserve Following Orbital Atherectomy and Percutaneous Revascularization in Severely Calcified Coronary Lesions
Brief Title: Coronary Flow Reserve Following Orbital Atherectomy
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN-0006-P
Record Dates: First submitted 2015-01-09; First posted 2015-01-15 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Stents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Enrolled Subjects: All subjects will receive Coronary Flow Reserve (CFR) measurements post successful orbital atherectomy treatment and stenting.
  Interventions: Device: Coronary Orbital Atherectomy plus Stenting

INTERVENTIONS:
Device: Coronary Orbital Atherectomy plus Stenting
  Other Names: DIAMONDBACK 360® Coronary Orbital Atherectomy System

SUMMARY:
The purpose of the study was to evaluate coronary artery flow reserve (CFR) following successful percutaneous coronary intervention (PCI) treatment of severely calcified coronary lesions by orbital atherectomy and stenting.

DETAILED DESCRIPTION:
This is an acute, observational, prospective, multi-center clinical study, evaluating coronary flow reserve (CFR) using the Volcano FloWire®. Subjects will be evaluated after treatment with orbital atherectomy and stenting of de-novo severely calcified lesions, due to coronary artery disease.

Subjects who undergo successful revascularization using the Diamondback 360® Coronary Orbital Atherectomy System (OAS) and stenting are eligible for enrollment. Coronary blood flow of enrolled subjects will be measured with the Volcano FloWire®, Doppler velocity data recorded intra-procedurally, and major adverse cardiac events (MACE) assessed at 24 hours or at discharge, whichever is earlier.

Determination of CFR by Doppler flow measurements can assess physiological changes in the distal vascular bed. The primary endpoint of this study will evaluate coronary flow reserve after successful treatment of severely calcified coronary lesions using OAS and stent deployment. The secondary endpoint will measure the occurrence of post-procedural Major Adverse Cardiac Events (MACE), including cardiac death, acute myocardial infarction (Q wave or non-Q wave), and target vessel revascularization.

ELIGIBILITY:
Subjects must meet all inclusion criteria and no exclusion criteria to be eligible to participate in the study.

Inclusion Criteria

1. Subjects must be at least 18 years of age.
2. Subjects must be scheduled for percutaneous coronary intervention involving stent deployment in de novo coronary lesions.
3. The target vessel must be a de-novo coronary artery with a severely calcified lesion.
4. The target vessel reference diameter must be ≥ 2.0mm and ≤ 4.0 mm.
5. The lesion length must not exceed 40 mm.
6. The target vessel must have a thrombolysis in myocardial infarction (TIMI) flow 3 at baseline.
7. The target lesion must have fluoroscopic, intravascular ultrasound (IVUS) or optical coherence tomograph (OCT) evidence of severe calcium deposit at the lesion site based on the protocol definition.
8. The lesion must be crossable with the ViperWire Advance® coronary guide wire.
9. Successful revascularization using OAS and stent deployment as demonstrated by no evidence of stent dissection and no more than 50% stenosis proximal to the stent.

Exclusion Criteria

1. Inability to understand the study or a history of non-compliance with medical advice.
2. Unwilling or unable to sign the informed consent form (ICF).
3. History of any cognitive or mental health status that would interfere with study participation.
4. Currently enrolled in any pre-approval investigational study. Note: This does not apply to long-term post-market studies unless these studies might clinically interfere with the current study endpoints.
5. Female subjects who are pregnant or planning to become pregnant within the study period.
6. Previous myocardial infarction of the target vessel.
7. Known sensitivity to contrast media, which cannot be adequately pre-medicated.
8. Diagnosed with chronic renal failure or has a serum creatinine level > 2.5 mg/dl.
9. History of a stroke or transient ischemic attack (TIA) within six (6) months of the procedure.
10. Active peptic ulcer or upper gastrointestinal (GI) bleeding within six (6) months of the procedure.
11. Wall motion abnormality in the intended vessel target zone.
12. Severe chronic obstructive pulmonary disease (COPD), asthma or current use of the medication: aminophylline.
13. 2nd or 3rd degree atrioventricular (AV) block.
14. Evidence of current left ventricular ejection fraction (LVEF) ≤45% (where current is defined as the latest LVEF measurement completed within the last 6 months).
15. New York Heart Association (NYHA) class III or IV heart failure.
16. Previous coronary artery bypass surgery.
17. Known allergy to atherectomy lubricant components such as soybean oil, egg yolk phospholipids, glycerin and sodium hydroxide.
18. Severe aortic stenosis.
19. Severe left ventricular hypertrophy.
20. Subject with angiographically confirmed evidence of more than 1 lesion requiring intervention.
21. Target vessel has other lesions with greater than 50% diameter stenosis based on visual estimate or on-line quantitative coronary analysis (QCA).
22. Target vessel has angiographically visible or suspected thrombus.
23. Target vessel has a stent from previous PCI unless:

    1. The stent was implanted greater than 30 days prior to the treatment, and
    2. The stent has no higher than 30% in-stent stenosis, and
    3. The stent is on a different branch than the target lesion.
24. Target vessel is excessively tortuous.
25. Target lesion is an ostial location (within 5 mm of ostium) or an unprotected left main lesion.
26. Target lesion is a bifurcation.
27. Target lesion has a ≥ 1.5 mm side branch.
28. Angiographic evidence of a dissection prior to initiation of orbital atherectomy device (OAD).
29. Angiographic evidence of MACE during procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been determined by their physician to require endovascular intervention for treatment of their CAD.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2015-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nabil Dib, MD, Principal Investigator — Dignity Health
Locations (3):
- United States (3):
  - Chandler Regional Medical Center and Mercy Gilbert Medical Center, Chandler, Arizona
  - Mercy Hospital, Coon Rapids, Minnesota
  - St. Francis Hospital, Roslyn, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Coronary Flow Reserve Assessment of Orbital Atherectomy: An Observational Pilot Study — https://www.scirp.org/journal/paperinformation.aspx?paperid=92106

RESULTS

PARTICIPANT FLOW:
Groups:
- Coronary Flow Reserve: Single arm - all enrolled subjects had successful coronary revascularization via orbital atherectomy and stenting.
Period: Overall Study
Arm/Group | Coronary Flow Reserve
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Coronary Flow Reserve
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.6 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 14
  American Indian or Alaska Native | 1

OUTCOME MEASURES:

1. Primary Outcome: Coronary Flow Reserve (CFR)
Description: CFR was measured after successful percutaneous coronary intervention (PCI) treatment of severely calcified coronary lesions. It was calculated from coronary blood flow velocity measurements, which were derived from Doppler-velocity wire data recorded in real time. The CFR formula utilized was APVp/APVb, where APVb is the average peak velocity at baseline and APVp is peak hyperemia.
Time Frame: Intra-procedurally following successful stent placement. Average procedure time 56 minutes.
Population: CFR is analyzed per protocol, which may require Doppler measurement in a control vessel in addition to the target vessel. Only subjects where this procedure is followed are included in the data set. The CFR formula is a ratio: APVp/APVb, where APV = average peak velocity (cm/sec). APVb = velocity at baseline and APVp = velocity at peak hyperemia.
Measure: Mean (Standard Deviation); unit: Ratio
Groups:
- All Eligible Subjects: All subjects whose Doppler flow measurements facilitated calculation of coronary flow reserve
Arm/Group | All Eligible Subjects
Number analyzed (Participants) | 8
Ratio | 2.23 (0.33)

2. Secondary Outcome: Major Adverse Cardiac Events (MACE)
Description: MACE: cardiac death, acute myocardial infarction (Q wave or non-Q wave), or target vessel revascularization.
Time Frame: At 24 hours or at time of hospital discharge, whichever occurred first
Population: MACE is evaluated per protocol, on subjects with successful PCI treatment of severely calcified coronary lesions
Measure: Number; unit: participants
Groups:
- All Enrolled Subjects: All subjects who have had successful revascularization by orbital atherectomy and stenting
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 15
participants | 0

ADVERSE EVENTS:
Time Frame: At 24 hours or at discharge, whichever was earlier.
Description: MACE defined as: Cardiac death, acute myocardial infarction (Q wave or non-Q wave), target vessel revascularization.
Arm/Group | All Enrolled Subjects
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled Subjects (N=15)
Cardiac Death (Cardiac disorders) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less